CLINICAL TRIAL: NCT02389777
Title: Effect of ACCS in UV-induced Inflammation
Brief Title: ST266 in UV-induced Inflammation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Noveome Biotherapeutics, formerly Stemnion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: ST-06-14
Record Dates: First submitted 2015-03-10; First posted 2015-03-17 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Skin Burns
MeSH Terms: conditions — Paresthesia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control UV burn (No Intervention): No treatment of the UV Light burn will be given
- ST266 treated UV burn immediately (Active Comparator): ST266 will be applied topically immediately by spray to the UV light burn wound
  Interventions: Biological: ST266 immediate
- ST266 treated UV burn delayed (Active Comparator): ST266 will be applied topically by spray to the UV light burn beginning 6 - 12 hours after the burn
  Interventions: Biological: ST266 delayed

INTERVENTIONS:
Biological: ST266 immediate — ST266 will be applied immediately to the UV light burn wound topically by spray twice per day
  Arms: ST266 treated UV burn immediately
Biological: ST266 delayed — ST266 will be applied to the UV light burn topically by spray twice per day beginning 6-12 hours after the burn
  Arms: ST266 treated UV burn delayed

SUMMARY:
This phase II clinical study will include fifteen healthy light skinned adult volunteers. At screening subjects will be given a sunburn test. This procedure involves exposing eight 1 square cm areas of skin over increasing doses of simulated solar radiation (SSR). SSR is delivered by a 1,000-Watt xenon arc lamp, which emits ultraviolet wavelengths from 290-400 nm, closely resembling natural sunlight. The Minimal Erythema Dose (MED) will be determined approximately 24 hours after initial exposure by using a chromometer. The MED is calculated by linear regression. Each test site is a one inch square area on the buttock or lower back. Sites 1, 2, 3, 4, 5 will be irradiated with 2 MED of SSR. Site 1 will not receive any ST266 treatment. Sites 2 and 3 will be treated with ST266 immediately after irradiation. 8-12 hours later or at bedtime, Sites 2,3,4,5 with ST266 at home. ST266 will also be applied 24 hours after SSR. Between 24-36 hours after SSR, subject returns to the Skin Study Center for Minolta chromometer assessment of erythema at all test sites, as well as for high resolution digital photography (Canfield). These assessments will be repeated at 48 hours and 72 hours post SSR. Data will be graphed to quantify rate of erythema resolution. Punch biopsies will be obtained at Site 1 (control) and Site 2 (SSR + immediate ST266 Rx). If a difference in erythema is observed between Site 1 and Site 4, a biopsy will also be obtained from Site 4 (SSR + delayed ST266 Rx). Biopsy samples will be tested using Reverse Transcriptase -Polymerase Chain Reaction (RT-PCR) and/or immunohistochemistry for markers of UV inflammation such as Interleukin (IL)-6, Tumor Necrosis Factor (TNF) -alpha, etc. Subjects will continue to apply the ST266 twice daily on Sites 3 and 5 until study visit 5. An additional normal control skin biopsy may be performed in a subset of volunteers (4-5) to serve as reference control for the tissue analysis.

DETAILED DESCRIPTION:
This phase II clinical study will include ten to fifteen healthy light skinned adult volunteers who will be recruited through Institutional Review Board (IRB)-approved advertising. At screening subjects will be given a sunburn test. This procedure involves exposing eight 1 square cm areas of skin over increasing doses of simulated solar radiation (SSR), while the rest of the body is draped. SSR is delivered by a 1,000-Watt xenon arc lamp, which emits ultraviolet wavelengths from 290-400 nm, closely resembling natural sunlight. The Minimal Erythema Dose (MED) will be determined approximately 24 hours after initial exposure by using a chromometer that records the values of redness associated with each 1 square cm area exposed to the SSR the previous day. Once the MED is calculated by linear regression, the actual UV exposure of test sites will be conducted. A test site consists of a one inch square area on the buttock or lower back. Sites 1, 2, 3, 4, 5 will be irradiated with 2 MED of SSR while the rest of the body is draped. Site 1 will not receive any ST266 treatment at all. Sites 2 and 3 will be treated by investigators with ST266 immediately after irradiation. 8-12 hours later or at bedtime, subject will treat Sites 2,3,4,5 with ST266 at home. ST266 application will also be done by subject on Sites 2,3,4,5 the next morning approximately 24 hours after SSR. Between 24-36 hours after SSR, subject returns to the Skin Study Center for Minolta chromometer assessment of erythema at all test sites, as well as for high resolution digital photography (Canfield). These assessments will be repeated at 48 hours and 72 hours post SSR and data will be graphed to quantify rate of erythema resolution. Punch biopsies will be obtained at Site 1 (control) and Site 2 (SSR + immediate ST266 Rx). If a difference in erythema is observed between Site 1 and Site 4 (i.e. if even the delayed treatment seems to effectively decrease inflammation), a biopsy will also be obtained from Site 4 (SSR + delayed ST266 Rx). These biopsy samples will be tested using RT-PCR and/or immunohistochemistry for markers of UV inflammation such as IL-6, TNF-alpha, etc. The test sites that have been biopsied will no longer undergo chromometer assessment post biopsy because the inflammation from the biopsy itself may confound the erythema readings. Meanwhile, subject will continue to apply the ST266 twice daily on Sites 3 and 5 until study visit 5. An additional normal control skin biopsy may be performed in a subset of volunteers (4-5) to serve as reference control for the tissue analysis. This will not be required of all volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 years or older
* Fitzpatrick Skin Type I-III
* In good general Adults health

Exclusion Criteria:

* Known history of photodermatosis or photosensitivity disorder such as systemic lupus or porphyria
* Tanning bed exposure within the last 4 weeks
* Current intake of known strong photosensitizers such as doxycycline/tetracycline family of antibiotics and thiazide diuretics
* Current intake of immunosuppressive drugs such as oral steroids.
* Cancer or known history of cancer within the last 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Erythema resolution | 3 days
  Erythema measured by Chromometer

SECONDARY OUTCOMES:
Skin punch biopsy | Baseline and end of study period (day 3)
  Punch biopsy will be assessed by RT-PCR and immunohistochemistry for markers of inflammation IL-6 and TNF-alpha

CONTACTS AND LOCATIONS:
Overall Officials: David L Steed, MD, Study Director — Noveome Biotherapeutics, formerly Stemnion; Elma D Baron, MD, Principal Investigator — Cae Western Reserve University

IPD SHARING:
Plan to Share IPD: No